CLINICAL TRIAL: NCT05218629
Title: Phase 2 Study of Anlotinib With PD-1 Inhibitor as Second Line Therapy in the Treatment of Metastatic Pancreatic Cancer
Brief Title: Anlotinib Plus PD-1 Inhibitor as 2nd-line Threapy in Patients With Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2022-01-18
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Overall Survival
MeSH Terms: interventions — anlotinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib， PD-1inhibitor (Experimental): Anlotinib 8-14 mg, oral, once a day for 14 days every 3 weeks. PD-1 inhibitor (Pembrolizumab) 200mg iv day1, every 3 weeks
  Interventions: Drug: Anlotinib, PD-1 inhibitor

INTERVENTIONS:
Drug: Anlotinib, PD-1 inhibitor — Anlotinib, 8-12 mg/day, orally, day 1-14; PD-1 inhibitor 200 mg iv, every 21 days one cycle

SUMMARY:
This research study is a Phase 2 clinical trial. It will test the efficiency and safety of an investigational drug of Anlotinib (a small molecular anti-VEGF TKI) with PD-1 inhibitor in second-line therapy with the goal of determining the OS of metastatic pancreatic adenocarcinoma. Subjects must have a stage 4 untreated metastatic pancreatic ductal cancer failed to first-line chemotherapy and meet all inclusion/exclusion criteria. Treatment consists of treatment with anlotinib 8-12 mg oral, day 1-14, and PD-1 inhibitor 200 mg iv, every 21 days each cycle. Treatment will be administered until untolerable toxicities or progression or subject death, or either the subject or sponsor discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically- or histologically-confirmed pancreatic adenocarcinoma or poorly differentiated pancreatic carcinoma that is metastatic to distant sites. • Other histologies such as neuroendocrine and acinar cell carcinoma are excluded. Enrolled patients are all failed to first-line chemotherapy • Patients are eligible if they received adjuvant treatment after surgical resection • Participants are required to have measurable disease (RECIST v1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan. See section 11 for the evaluation of measurable disease. • Participants enrolled must have disease that is accessible for tumor biopsies and must agree to a pre-treatment tumor biopsy. • Age ≥ 18 years. Because no dosing or adverse event data are currently available in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials. • ECOG performance status ≤2 (see Appendix A) • Patients must have completed any major surgery or open biopsy ≥4 weeks from start of treatment. • Participants must have adequate organ and marrow function as defined below: o Absolute neutrophil count ≥1,500/mcL o Platelets ≥100,000/mcL o Total bilirubin ≤1.5 × institutional upper limit of normal o AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal o Creatinine ≤1.5 × institutional upper limit of normal OR o Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × upper limit of normal. • Negative serum pregnancy test for women of childbearing potential. • Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents. • Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Screening for brain metastases with head imaging is not required. • History of allergic reactions attributed to compounds of similar chemical or biologic composition to above drugs or other agents used in study. • History of prior or current synchronous malignancy, except: o Malignancy that was treated with curative intent and for which there has been no known active disease for >3 years prior to enrollment • Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, NYHA class III/IV congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The overall survival in this population of patients | 24 months
  The overall survival of the enrolled patients from start the combination treatment of anlotinib and PD-1 inhibitor

SECONDARY OUTCOMES:
The progression free survival in this population of patients | 24 months
  The progression free survival of the enrolled patients from start the combination treatment with anlotinib and PD-1 inhibitor
The response rate in this population of patients | Up to 48 months
  Number of participants with clinical response assessed by RECIST 1.1 criteria on imaging every 4 weeks with the combination of anlotinib and PD-1 inhibitor

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao central Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR